CLINICAL TRIAL: NCT07079514
Title: Role of Magnesium Sulphate Versus Placebo on Hemodynamic Changes During Pneumoperitoneum During Laparoscopic Procedures
Brief Title: Effect of Magnesium Sulfate on Hemodynamics on Laparoscopic Cholecystectomy Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Ziauddin University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 8840724RHANE
Record Dates: First submitted 2025-07-02; First posted 2025-07-23 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-06

CONDITIONS: Hemodynamics Instability; Pain After Surgery; PONV in Laparoscopic Cholocystectomies
Keywords: Pneumoperitoneum; Hemodynamics; Magnesium Sulfate; Pain; PONV
MeSH Terms: conditions — Pneumoperitoneum; Pain; Postoperative Nausea and Vomiting | interventions — Magnesium; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group A (Placebo Comparator): 100ml normal saline is used as placebo
  Interventions: Drug: Placebo
- groupB (Active Comparator): 3g magnesium sulphate
  Interventions: Drug: Magnesium

INTERVENTIONS:
Drug: Placebo — normal saline in 100ml piggy bag
  Arms: group A
Drug: Magnesium — Magnesium Sulphate will be given as doses of 20-50mg/kg in 2 -3 minutes. In order to standardize the dose in every patient we will be using 3g
  Other Names: MgSo4; Magnesium sulphate
  Arms: groupB

SUMMARY:
The goal of this triple blinded randomized control trial is to compare the effect of magnesium sulphate on the hemodynamic response during pneumoperitoneum creation, along with its impact on postoperative pain, opioid consumption, and post operative nausea vomiting (PONV) in ASA I to III patients undergoing laparoscopic cholecystectomy The main question[s] it aims to answer is whether the agent Magnesium Sulphate will blunt the increase in the hemodynamic response during peritoneal insufflation, and will it decrease post operative opioids consumption and prevent nausea vomiting in patients undergoing laparoscopic surgeries.

30 were given placebo and 30 were introduced with magnesium sulphate (3mg) 5 mins before insufflation. The hemodynamic such as, mean arterial pressure (MAP,) systolic (SBP) and diastolic blood pressures (DBP), heart rate (HR) were recorded pre operatively and intraoperatively with intervals of 5mins. Pain score was recorded by VAS scaling and post operative nausea vomiting (PONV) with Yes and No in post operative anesthesia unit (PACU) period.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85
* Gender: Male /Female
* ASA status I/II/III
* Patients undergoing elective Laparoscopic cholecystectomy

Exclusion Criteria:

* Known Hypermagnesemia
* Known allergy to Magnesium
* Any degree of Heart Block
* Patients on Calcium Channel Blockers
* Known CKD/AKI

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-04-21 (Actual); Study Completion 2025-04-21 (Actual)

PRIMARY OUTCOMES:
Changes in Mean arterial pressures (MAP), Systolic blood pressures (SBP), Diastolic blood pressures (DBP) | 6 months
  Laparoscopic surgeries, such as cholecystectomy, require CO₂ insufflation to create pneumoperitoneum, which leads to increased sympathetic activity, elevated blood pressure
Changes in Heart Rate (HR) | 6 months
  Laparoscopic surgeries, such as cholecystectomy, require CO₂ insufflation to create pneumoperitoneum

SECONDARY OUTCOMES:
Pain Scores on the Visual Analog SCALE | 6 months
  magnesium sulfate acts on NMDA receptor and has non opioid pain relieving properties hence we are going to assess whether there's a decrease in post operative pain

OTHER OUTCOMES:
YES/NO questionnaire for Post operative nausea vomiting | 6 months
  post operative nausea vomiting assessment will through yes or no questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Dr Asma A Salam, MBBS, FCPS, Study Chair — Dr Ziauddin Hospital
Locations (1):
- Dr Ziauddin Hospital, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
written consent, demographics, co-morbids, hemodynamic parameters of each patients. duration of surgery, total anesthesia duration, time for which pneumoperitoneum was created.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: 6 months

REFERENCES:
- [Result] Shafiq T, Rana MA, Nisar A. Comparison of Hemodynamic Response after Pneumoperitoneum with Versus without Pre-Emptive Magnesium Sulphate in Patients Undergoing Laparoscopic Cholecystectomy. Pakistan Journal of Medical & Health Sciences. 2022 Apr 12;16(03):267
- [Result] Maya G, Ramya N, Anzar S, et al. Effect of magnesium sulfate in attenuating arterial blood pressure in elective laparoscopic abdominal surgeries. J. Evolution Med. Dent. Sci. 2017;6(33):2680-2683, DOI: 10.14260/Jemds/2017/578
- [Result] Zareen A, Gardazi SFA, Anwar MH, Zaheer J. Effects of IV Magnesium Sulphate on Hemodynamic Response to Pneumoperitoneum in Laparoscopic Cholecystectomy; A randomized control. Ann Pak Inst Med Sci. 2021; 17(2):82-85. doi. 10.48036/apims.v17i2.539
- [Result] Murumu DP, Mishra M, Singh AK, Mathur SK. Effect of Magnesium Sulphate on Intra Operative Anesthetic Requirements and Post Operative Analgesia in Plastic Surgery Patients. Int J Anesth Res. 2021 Nov 29;9(03):662-7.
- [Result] Tramer MR, Glynn CJ. An evaluation of a single dose of magnesium to supplement analgesia after ambulatory surgery: randomized controlled trial. Anesth Analg. 2007 Jun;104(6):1374-9, table of contents. doi: 10.1213/01.ane.0000263416.14948.dc. PMID 17513629
- [Result] Paul S, Biswas P, Bhattacharjee DP, Sengupta J. Effects of magnesium sulfate on hemodynamic response to carbon dioxide pneumoperitoneum in patients undergoing laparoscopic cholecystectomy. Anesth Essays Res. 2013 May-Aug;7(2):228-31. doi: 10.4103/0259-1162.118970. PMID 25885838
- [Result] Jee D, Lee D, Yun S, Lee C. Magnesium sulphate attenuates arterial pressure increase during laparoscopic cholecystectomy. Br J Anaesth. 2009 Oct;103(4):484-9. doi: 10.1093/bja/aep196. Epub 2009 Jul 17. PMID 19617379
- [Result] Do SH. Magnesium: a versatile drug for anesthesiologists. Korean J Anesthesiol. 2013 Jul;65(1):4-8. doi: 10.4097/kjae.2013.65.1.4. Epub 2013 Jul 19. PMID 23904932
- [Result] Tripathi DC, Shah KS, Dubey SR, Doshi SM, Raval PV. Hemodynamic stress response during laparoscopic cholecystectomy: Effect of two different doses of intravenous clonidine premedication. J Anaesthesiol Clin Pharmacol. 2011 Oct;27(4):475-80. doi: 10.4103/0970-9185.86586. PMID 22096279
- [Result] Tan W, Qian DC, Zheng MM, Lu X, Han Y, Qi DY. Effects of different doses of magnesium sulfate on pneumoperitoneum-related hemodynamic changes in patients undergoing gastrointestinal laparoscopy: a randomized, double-blind, controlled trial. BMC Anesthesiol. 2019 Dec 20;19(1):237. doi: 10.1186/s12871-019-0886-4. PMID 31862004
- [Result] El Mourad MB, Arafa SK. Effect of intravenous versus intraperitoneal magnesium sulfate on hemodynamic parameters and postoperative analgesia during laparoscopic sleeve gastrectomy-A prospective randomized study. J Anaesthesiol Clin Pharmacol. 2019 Apr-Jun;35(2):242-247. doi: 10.4103/joacp.JOACP_208_18. PMID 31303716
- See also: Effectiveness of intravenous magnesium sulfate to attenuate hemodynamic changes in laparoscopic surgery: a systematic review and meta-analysis — https://pubmed.ncbi.nlm.nih.gov/33074990/